CLINICAL TRIAL: NCT00773162
Title: A Single-center, Randomized, Double-blind, Phase III Comparison of the Efficacy and Safety of Quetiapine Fumarate (Oral Extended Release Tablets) to Placebo in Social Phobia Patients and Changes in Their Vasodilatory Response to Methyl-Nicotinate
Brief Title: Flushing in Social Anxiety Disorder on Seroquel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: START Clinic for Mood and Anxiety Disorders (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Martin A. Katzman, Principal Investigator, START Clinic for Mood and Anxiety Disorders
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AzSeroSP
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Quetiapine Fumarate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Sugar Pill
- 2 (Active Comparator)
  Interventions: Drug: Seroquel

INTERVENTIONS:
Drug: Seroquel — seroquel XR- oral extended release tablets, 50mg - 300mg, 16 weeks
  Other Names: Quetiapine
  Arms: 2
Drug: Sugar Pill — Sugar pill to match seroquel
  Arms: 1

SUMMARY:
To add to our understanding of the relationship between blushing, symptom severity and potential mechanisms that underlie blushing in patients with Social Phobia (SP), the investigators propose comparing SP patients' vascular responses to topical m-N pre and post treatment with Seroquel or placebo.

Atypical antipsychotics such as seroquel have been used successfully as adjunctive treatments in other anxiety disorders, including PTSD (Labatte, 2001; Krashin & Oates, 1999; McDougle et al., 2000; Pfanner et al., 2000; Bogetto et al., 2000) and Generalized Anxiety Disorder (Katzman et al., 2005). Responses to the blushing exposure will be assessed prior to and following treatment with seroquel or placebo and at one month following intervention. Levels of prostaglandin will be compared between groups and will also be correlated with symptom severity in the clinical groups.

The objective of this randomized, double blind flexible -dose study will be to evaluate the efficacy , safety and tolerability of seroquel SR 50mg to 800mg and placebo in outpatient subjects diagnosed with SP. The study will begin with a single week of Seroquel 50mg or placebo. Subsequently, tablets will be administered by the investigator in a flexible dose fashion during the visits. Patients will be followed up weekly (biweekly after week 6) and at the clinician's discretion. After the fist week the patients' dosage will be increased up to a maximum of 800 mg daily with expected average dose of 300mg dail. This dose will remain fixed after 8 weeks of treatment until week 16.

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided signed informed consent prior to any study-related procedures
* Outpatient male or female aged 18-65 (inclusive).
* Patients with a primary diagnosis of Social Phobia to DSM IV (300.23) criteria (diagnosis to be made using the MINI International Neuropsychiatric Interview (MINI).
* Score of > 60 on the LSAS.
* On the basis of a physical examination, medical history and basic laboratory screening, the patient is, in the investigator's opinion, in suitable condition.

Exclusion Criteria:

* Pregnancy or lactation
* Any DSM-IV Axis I disorder not defined in the inclusion criteria
* Patients who, in the opinion of the investigator, pose an immediate risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following P450 3A4 inhibitors in the 14 days preceding enrollment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine, and saquinavir.
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids.
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization
* Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by the DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
* Positive drug screen result at screening visit and if clinically relevant judged by the investigator
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illnesses (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning or conduct of the study
* Previous enrollment or randomization of treatment in the present study
* Participation in another drug trail within 4 weeks prior enrollment into this study or longer in accordance with local requirements
* Continuation or commencement of formal psychotherapy
* Current use of or commencement of antidepressant and anxiolytic medications
* Patients, who have been on an antidepressant or other anxiolytic prior to the study, will have discontinues these more than two weeks prior to entry into the study. Those who have been on fluoxetine, will have been off for at least five weeks.
* Patients, who have been on a herbal or alternative treatment judged to be potentially anxiolytic or with psychobiological activity, will have terminated usage of the agent more than two weeks prior to entering the study
* Previous reactions to Niacin administration
* Use of a non-steroidal anti-inflammatory
* Any psychotic disorder
* Eating disorder as defined in the DSM IV
* Mental retardation or other cognitive disorder
* Laboratory values at screening or in medical history that may be considered through clinical interpretation to be significant
* Serious illness: Liver or renal insufficiency, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic or metabolic disturbance
* An absolute neutrophil count (ANC) of <1.5 x 109 per liter.
* Unstable Diabetes Mellitus/HbA1c

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in intensity of the vasodilatory response to 10 mM topical m-N over 16 weeks. | 20 weeks

SECONDARY OUTCOMES:
Mean change from baseline on the HAM-A, CGI, SF-36, LSAS, SPIN, SIAS, SPS, ASI, BAI, BDI, SHEEHAN, EUROQUEL, BIS/BAS, PSWQ, IUS | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Katzman, MD, Principal Investigator — START Clinic for Mood and Anxiety Disorders
Locations (1):
- START Clinic for the Mood and Anxiety Disorders, Toronto, Ontario, Canada